CLINICAL TRIAL: NCT01187875
Title: Satiety Response of Resistant Starches
Brief Title: Resistant Starch and Satiety
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 806M37445
Record Dates: First submitted 2010-06-21; First posted 2010-08-24 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Adults
Keywords: satiety, dietary fiber

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Dextrin Control
  Interventions: Dietary Supplement: Placebo- Fiber free control
- Hi-maize resistant starch 9g (Experimental): Hi-maize resistant starch 9g
  Interventions: Dietary Supplement: Hi-maize resistant starch 9g
- Novalose 330 resistant starch 9g (Experimental): Novalose 330 resistant starch 9g
  Interventions: Dietary Supplement: Novalose 330 resistant starch 9g
- 4.5g Hi-maize and 4.5g Novalose 330 (Experimental): 4.5g Hi-maize and 4.5g Novalose 330
  Interventions: Dietary Supplement: 4.5g Hi-maize resistant starch and 4.5g Novalose 330

INTERVENTIONS:
Dietary Supplement: Placebo- Fiber free control — Dextrin control administered in a muffin treatment.
  Arms: Control
Dietary Supplement: Hi-maize resistant starch 9g — 9g Hi-maize resistant starch administered in a muffin treatment.
  Arms: Hi-maize resistant starch 9g
Dietary Supplement: Novalose 330 resistant starch 9g — 9g Novalose 330 resistant starch administered in a muffin treatment.
  Arms: Novalose 330 resistant starch 9g
Dietary Supplement: 4.5g Hi-maize resistant starch and 4.5g Novalose 330 — 4.5g Hi-maize and 4.5g Novalose 330 in a muffin treatment.
  Arms: 4.5g Hi-maize and 4.5g Novalose 330

SUMMARY:
Dietary fiber consumption may contribute to weight regulation by improving satiety. In an earlier study the investigators found that a muffin containing resistant starch was more effective than other fibers in altering satiety. The objective of this study is to determine if 2 resistant starches consumed in muffins alter satiety and whether a mixture of resistant starches is more effective than either alone in enhancing satiety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-64 years
* Non-smoking
* Not taking medication
* Non dieting (weight stable in prior 3 months)
* BMI 18-27
* English literacy

Exclusion Criteria:

* Do not regularly consume breakfast
* Food allergies to ingredients found in the study products
* BMI <18 or >27
* Diagnosed cardiovascular disease, renal disease, hepatic disease, or diabetes mellitus
* Cancer in previous 5 years
* Any gastrointestinal disease or condition
* Recent bacterial infection (< 3months)
* Recent or concurrent participation in an intervention research study
* History of drug or alcohol abuse in prior 6 months
* Use of lipid lowering, anti-hypertensive, or anti-inflammatory steroid medication
* Eating disorder
* Vegetarians
* People who eat more than approximately 15 grams of fiber per day
* Women who are pregnant or lactating
* Women with irregular menstrual cycles

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Satiety response using visual analogue scales | 0 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 15 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 30 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 45 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 60 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 90 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 120 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 180 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).
Satiety response using VAS | 240 minutes postprandially
  Satiety response was measured using subjective perceptions of hunger, fullness, satisfaction, and prospective food intake evaluated by previously validated visual analogue scales (VAS).

SECONDARY OUTCOMES:
Ad libitum food intake | 240 minutes postprandially and over 24 hours
Breath hydrogen response | 0, 240 minutes
Gastrointestinal tolerance using visual analogue scales (VAS) | 24 hours
  Subjective ratings of bloating, stool consistency, and flatulence on VAS. A stool count was also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Saint Paul, Minnesota, United States